CLINICAL TRIAL: NCT05837455
Title: NeoTAILOR: A Phase II Biomarker-directed Approach to Guide Neoadjuvant Therapy for Patients With Stage II/III ER-positive, HER2-negative Breast Cancer
Brief Title: NeoTAILOR: ABiomarker-directed Approach to Guide Neoadjuvant Therapy for Patients With Stage II/III ER-positive, HER2-negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Swim Across America (Other); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202305007
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Cancer of the Breast
Keywords: breast cancer; postmenopausal women; Ki67; PAM50 subtype; breast cancer disparities
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Low-risk group (Experimental): * Baseline breast MRI and research specimen collection prior to the start of treatment with standard of care anastrozole. All patients will have one 28-day cycle of anastrozole, followed by determination of breast cancer risk category by incorporating results from baseline Ki67, Oncotype DX RS, and molecular intrinsic subtype by PAM50.
  * An additional blood draw for research purposes at Week 4 (no breast tumor biopsy at this time point) and continue to receive 5 additional 28-day cycles of anastrozole.
  * After completion of ~6 months of neoadjuvant treatment, will undergo post-treatment breast MRI followed by standard of care surgery.
  Interventions: Device: VENTANA MIB-1 Ki67 assay; Device: Oncotype DX® Recurrence Score; Device: PAM50-based Prosigna breast cancer gene signature assay; Drug: Anastrozole
- High-risk endocrine-sensitive group (Experimental): * Baseline breast MRI and research specimen collection prior to the start of treatment with standard of care anastrozole. All patients will have one 28-day cycle of anastrozole, followed by determination of breast cancer risk category by incorporating results from baseline Ki67, Oncotype DX RS, and molecular intrinsic subtype by PAM50.
  * An additional blood draw and breast tumor tissue collection at Week 4 to assess Ki67. Patients with Week 4 Ki67 ≤10% (the high-risk endocrine-sensitive group) will continue to receive 5 additional 28-day cycles of anastrozole.
  * After completion of ~6 months of neoadjuvant treatment, will undergo post-treatment breast MRI followed by standard of care surgery.
  Interventions: Device: VENTANA MIB-1 Ki67 assay; Device: Oncotype DX® Recurrence Score; Device: PAM50-based Prosigna breast cancer gene signature assay; Drug: Anastrozole
- High-risk endocrine-resistant group (Experimental): * Baseline breast MRI and research specimen collection prior to the start of treatment with standard of care anastrozole. All patients will have one 28-day cycle of anastrozole, followed by determination of breast cancer risk category by incorporating results from baseline Ki67, Oncotype DX RS, and molecular intrinsic subtype by PAM50.
  * An additional blood draw and breast tumor tissue collection at Week 4 to assess Ki67. Patients with Week 4 Ki67 >10% (the high-risk endocrine-resistant group) will receive escalated therapy with ~5-6 additional months of standard of care chemotherapy (combination anthracycline- and/or taxane-based at the discretion of their physician).
  * After completion of ~6 months of neoadjuvant treatment, will undergo post-treatment breast MRI followed by standard of care surgery.
  Interventions: Device: VENTANA MIB-1 Ki67 assay; Device: Oncotype DX® Recurrence Score; Device: PAM50-based Prosigna breast cancer gene signature assay; Drug: Combination anthracycline and/or taxane based treatment

INTERVENTIONS:
Device: VENTANA MIB-1 Ki67 assay — Ki67 scoring determination (standard of care) utilizing the Ki67 MIB-1 assay (clone 30-9) (VENTANA) will be performed at baseline, Week 4 (+/- 14 days - high-risk group only), and at time of surgery in accordance with the International Ki67 in Breast Cancer Working Group guidelines.
Device: Oncotype DX® Recurrence Score — Oncotype DX® Recurrence Score (RS) testing - assessing expression of 21 genes including 16 cancer-related genes and 5 reference genes - will be performed as standard of care in a central laboratory (Exact Sciences) on RNA extracted from formalin-fixed paraffin-embedded core-biopsy samples.
Device: PAM50-based Prosigna breast cancer gene signature assay — This PAM50-based Prosigna breast cancer gene signature assay for intrinsic molecular subtype determination will be performed on formalin-fixed, paraffin-embedded (FFPE) core-biopsy samples.
Drug: Anastrozole — Standard of care
  Arms: High-risk endocrine-sensitive group; Low-risk group
Drug: Combination anthracycline and/or taxane based treatment — Standard of care
  Arms: High-risk endocrine-resistant group

SUMMARY:
This study aims to utilize a novel biomarker-driven approach to guide neoadjuvant treatment selection. It is the hypothesis that this will improve clinical response for postmenopausal women with clinical stage II/III ER-positive, HER2-negative breast cancer and identify those who may not require neoadjuvant chemotherapy, with a primary focus on outcomes in Black patients.

DETAILED DESCRIPTION:
Risk category is defined as follows:

* Low risk:

  * Baseline Ki67 ≤ 10% (OR)
  * Luminal A molecular intrinsic subtype by PAM50
* High risk:

  * Non-Luminal A molecular intrinsic subtype by PAM50 (OR)
  * In cases of non-diagnostic PAM50 molecular intrinsic subtype, patients will enroll in the high-risk group and undergo Week 4 tumor biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed newly diagnosed clinical stage II or III (by AJCC 8th edition - at least T2, any N, M0 or if N1+ then any T) ER-positive (ER > 10%), any PR, and HER2-negative breast cancer with complete surgical excision of the breast cancer after neoadjuvant therapy as the treatment goal.

  * HER2 negative must be assessed by FISH or IHC staining 0 or 1+ according to ASCO/CAP guidelines.
* A palpable mass is not required; however, tumor size must be either:

  * ≥2 cm in one dimension by clinical or radiographic examination (WHO criteria), if clinically axillary lymph node negative OR
  * Measureable (≥10 mm) by modified RECIST v1.1 for breast MRI (see Section 9.0), if histologically confirmed resectable locoregional nodal involvement.
* ECOG performance status 0 or 1.
* Eligible to receive neoadjuvant aromatase inhibitor, as per treating physician.
* Eligible to receive neoadjuvant standard of care anthracycline- and/or taxane-based chemotherapy regimen, as per treating physician.
* Able to tolerate breast MRI with intravenous contrast administration. Must be able to complete the applicable MRI screening evaluation form.
* Adequate bone marrow and organ function, as determined by the treating physician.
* Known history of hepatitis C virus (HCV) infection is permissible provided the patient has been treated and cured.
* At least 18 years of age.
* Postmenopausal status, defined as one of the following:

  * Age ≥ 60 years
  * Age < 60 with intact uterus and amenorrhea for 12 consecutive months or more
  * Status post bilateral oophorectomy, total hysterectomy
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable), and willing and able to comply with scheduled visits and treatment schedule.

Exclusion Criteria:

* Inflammatory breast cancer (cT4d disease as per AJCC 8th edition).
* Locally recurrent or metastatic disease (cM1 disease as per AJCC 8th edition).
* Bilateral breast cancer.
* Prior systemic therapy for the indexed breast cancer.
* Pre-existing Grade ≥2 neuropathy.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* A history of other malignancy ≤5 years prior to the indexed breast cancer diagnosis with the following exceptions:

  * Basal cell or squamous cell carcinoma of the skin which were treated with local resection only
  * Adequately treated carcinoma in situ of the cervix.
  * Prior or concurrent malignancy whose natural history or treatment will not interfere with the safety or efficacy assessments of the indexed breast cancer. In this event, review and approval by the study PI is required.
* Concurrent participation in any investigational therapeutic trial for treatment of breast cancer.
* Known HIV positivity that in the judgement of the treating physician would impact safety of chemotherapy receipt.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to anastrozole, taxanes (paclitaxel or nab-paclitaxel), anthracyclines (doxorubicin or epirubicin) or cyclophosphamide.
* Evidence of uncontrolled ongoing or active infection, requiring parenteral anti-bacterial, anti-viral, or anti-fungal therapy ≤ 7 days prior to administration of study treatment. Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible.
* Any uncontrolled medical condition that in the opinion of the Investigator would pose a risk to participant safety or interfere with study participation or interpretation of individual participant results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by breast MRI in the combined low-risk plus high-risk endocrine-sensitive groups (pooled endocrine therapy-responders) | Through completion of treatment (estimated to be 6 months)
  * ORR is defined as patients achieving clinical complete response (CR) or partial response (PR) according to RECIST v1.1.
  * Complete Response (CR): disappearance of all target and non-target lesions. Residual lesions thought to be non-malignant should be further investigated before CR can be accepted.
  * Partial Response (PR): ≥30% decrease in the sum of measures of target lesions, taking as reference the baseline sum of diameters. Non-target lesions must be non-PD.

SECONDARY OUTCOMES:
Breast conservation surgery (BCS) conversion rate by cohort and treatment assignment | Through completion of surgery (estimated to be 6 months)
Proportion of patients who will require oncoplastic breast reduction surgery before and after neoadjuvant treatment | Through completion of surgery (estimated to be 6 months)
Objective response rate (ORR) by breast MRI in the high-risk endocrine-sensitive group | Through completion of treatment (estimated to be 6 months)
  * ORR is defined as patients achieving clinical complete response (CR) or partial response (PR) according to modified RECIST v1.1.
  * Complete Response (CR): disappearance of all target and non-target lesions. Residual lesions thought to be non-malignant should be further investigated before CR can be accepted.
  * Partial Response (PR): ≥30% decrease in the sum of measures of target lesions, taking as reference the baseline sum of diameters. Non-target lesions must be non-PD.
Objective response rate (ORR) by breast MRI in the high-risk endocrine-resistant group (high risk patients with week 4 Ki67 > 10% post anastrozole) | Through completion of treatment (estimated to be 6 months)
  * ORR is defined as patients achieving clinical complete response (CR) or partial response (PR) according to modified RECIST v1.1.
  * Complete Response (CR): disappearance of all target and non-target lesions. Residual lesions thought to be non-malignant should be further investigated before CR can be accepted.
  * Partial Response (PR): ≥30% decrease in the sum of measures of target lesions, taking as reference the baseline sum of diameters. Non-target lesions must be non-PD.

CONTACTS AND LOCATIONS:
Overall Officials: Nusayba Bagegni, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu